CLINICAL TRIAL: NCT07154446
Title: Dynastat vs. Parestat for Postoperative Analgesia in Breast Surgery: A Non-Inferiority Randomised Controlled Trial
Brief Title: Study Comparing Dynastat and Parestat Pain Relief Medications for Patients After Breast Surgery
Acronym: PANDA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Ahmad Fariz Bin Elias, Dr, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202557-15040
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Exicision Biopsy
Keywords: Randomised control trial; parecoxib; Breast excision biopsy
MeSH Terms: interventions — parecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parestat Group, Parestat(generic parecoxib) (Experimental): Patients receiving IV Parestat 40mg (generic Parecoxib) will have it administered by an anaesthesiologist after the induction of general anaesthesia and before the surgeon makes the skin incision.
  Interventions: Drug: Parestat(generic parecoxib)
- Dynastat group, Dynastat(Original Parecoxib) (Active Comparator): Patients receiving IV Dynastat 40mg (original Parecoxib) will have it administered by an anaesthesiologist after the induction of general anaesthesia and before the surgeon makes the skin incision.
  Interventions: Drug: Dynastat (original Parecoxib)

INTERVENTIONS:
Drug: Parestat(generic parecoxib) — This arm will receive IV Parestat 40mg during surgery
  Arms: Parestat Group, Parestat(generic parecoxib)
Drug: Dynastat (original Parecoxib) — This arm will receive IV Dynastat 40mg during surgery
  Arms: Dynastat group, Dynastat(Original Parecoxib)

SUMMARY:
The goal of this clinical trial is to learn if generic parecoxib (Parestat) works as well as the original drug (Dynastat) for treating pain after breast surgery. It will also learn about the safety of both drugs. The main questions it aims to answer are:

* Does Parestat provide pain relief that is not inferior to the pain relief provided by Dynastat?
* What medical problems (adverse events) do participants have when taking Parestat compared to Dynastat? Researchers will compare Parestat to Dynastat to see if the generic version also works to treat postoperative pain.

Participants will:

* Be randomly assigned to receive either Dynastat or Parestat during their surgery.
* Have their pain level assessed using the Visual Analog Scale (VAS) upon arrival in the recovery bay, 6 and 24 hours after surgery.
* Be monitored for common side effects like nausea, vomiting, and changes in blood pressure for 24 hours.

DETAILED DESCRIPTION:
The goal of this clinical trial is to determine whether generic parecoxib (Parestat) is as effective as the original parecoxib (Dynastat) for treating pain following breast surgery. The trial will also assess the safety of both medications. The main questions it aims to answer are:

1. Does generic parecoxib (Parestat) provide the same level of pain relief as original parecoxib (Dynastat) after breast biopsy surgery?
2. What side effects do participants experience when taking either medication?

Researchers will compare Parestat to Dynastat to see if the generic version is equally effective for managing postoperative pain.

Participants in the study will:

* Receive either Parestat or Dynastat during their breast excision biopsy surgery.
* Have their pain levels measured using a pain scale at three time points: in the recovery room, before transferring to the ward, and 24 hours after surgery.
* Be monitored for side effects such as nausea, changes in blood pressure, swelling, and other adverse reactions for 24 hours.
* Be kept unaware of which medication they received (double-blind study design).

The study will involve 60 adult women undergoing elective breast biopsy surgery, with 30 participants in each treatment group.t group.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 18 years or older. Patients scheduled for elective excision biopsy of the breast. Patients with an American Society of Anesthesiologists (ASA) physical status classification of I or II.

Patients who can understand and provide written informed consent.

Exclusion Criteria:

Patients with a known allergy or contraindication to parecoxib or any of its excipients.

Patients with a history of severe gastrointestinal bleeding, ulceration, or perforation.

Patients with a history of significant cardiovascular disease (e.g., unstable angina, recent myocardial infarction, stroke).

Patients with uncontrolled hypertension. Patients with severe renal impairment (creatinine clearance < 30 mL/min). Patients with severe hepatic impairment (Child-Pugh Class C). Patients who are pregnant or breastfeeding. Patients taking medications that are contraindicated with parecoxib (refer to drug interaction section).

Patients with a history of bronchospasm, acute rhinitis, nasal polyps, angioedema, urticaria, or other allergic-type reactions after taking aspirin or other NSAIDs.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female, as identified by a Malaysian identity card or passport
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Pain Score | 24 hours after surgery completed
  Each participant's pain score will be assessed using the Numeric Rating Scale (NRS) at three time points: upon arrival in the recovery bay, before discharge from the recovery bay, and 24 hours postoperatively.
  The NRS ranges 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Highest score reflect worst outcome

SECONDARY OUTCOMES:
Adverse events | 24 hours after completion of surgery
  To detect and compare the incidence of common adverse events between the two groups, specifically:
  * Nausea and vomiting, constipation
  * Changes in blood pressure, differences 20% from baseline (increase or decrease)
  * Edema
  * Pruritus
  * Gastritis
  * Bronchospasm

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Fariz Elias, Principal Investigator — Universiti Malaya

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices), will be made available beginning 9 months and ending 36 months following article publication to researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, ICF
Time Frame: January 2026 until january 2027
Access Criteria: Data will be made available to qualified researchers affiliated with recognized academic institutions, government agencies, or non-profit organizations who provide a methodologically sound proposal
URL: https://redcap.um.edu.my/index.php